CLINICAL TRIAL: NCT05614921
Title: Ultrasound Guided External Oblique Intercostal Plane Block vs. Wound Infiltration for Laparoscopic Sleeve Gastrectomy: Prospective Randomized Study
Brief Title: External Oblique Intercostal Plane Block vs. Wound Infiltration for Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: Erzurum City Hospital (Other); Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: atauniobesity
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External oblique intercostal plane block (Active Comparator): Ultrasound-guided External oblique intercostal plane block before surgery
  Interventions: Other: ultrasound guided external oblique intercostal plane block
- Wound infiltration (Active Comparator): Wound infiltration to trocar sites before surgery
  Interventions: Other: Wound infiltration

INTERVENTIONS:
Other: ultrasound guided external oblique intercostal plane block — ultrasound guided external oblique intercostal plane block 30 ml local anesthetic each side
  Arms: External oblique intercostal plane block
Other: Wound infiltration — 5 ml local anesthetic for each trocar side
  Arms: Wound infiltration

SUMMARY:
The morbidity and mortality associated with being overweight or obese have been known to the medical profession since Hippocrates, more than 2500 years ago.

Pain that develops following bariatric surgery may prolong recovery time. Most morbidly obese patients have obstructive sleep apnea and cardiac comorbidities. In these patients, prolonged postoperative pain may cause early ambulation and delay performing deep breathing exercises.

Using regional anesthetic techniques results in less opioid use and better pain management. External oblique internal costal block; It is a new block that provides dermatomal sensory blockage involving T6-T10 in the anterior axillary line and T6-T9 in the midline. It can be used as part of multimodal analgesia in laparoscopic cases.

There is no study in the literature regarding the use of external oblique plane block in bariatric surgery yet.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-III patients
* Laparoscopic Obesity surgery

Exclusion Criteria:

* Chronic pain bleeding disorders renal or hepatic insufficiency patients on chronic non-steroidal anti-inflammatory medications emergency cases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | first 24 hours
  First 24 hours total fentanyl consumption with patient controlled analgesia

SECONDARY OUTCOMES:
Visual analog pain score | postextubation 0-24 hours
  Post operative pain will be evaluated with a Visual Analogue Scale (VAS) score of 0-10 (0= no pain and 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] White L, Ji A. External oblique intercostal plane block for upper abdominal surgery: use in obese patients. Br J Anaesth. 2022 May;128(5):e295-e297. doi: 10.1016/j.bja.2022.02.011. Epub 2022 Mar 3. No abstract available. PMID 35249704
- [Background] Cosarcan SK, Yavuz Y, Dogan AT, Ercelen O. Can Postoperative Pain Be Prevented in Bariatric Surgery? Efficacy and Usability of Fascial Plane Blocks: a Retrospective Clinical Study. Obes Surg. 2022 Sep;32(9):2921-2929. doi: 10.1007/s11695-022-06184-9. Epub 2022 Jul 1. PMID 35776242